CLINICAL TRIAL: NCT03168347
Title: Assessing Patient Confidence in Biologic Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB00043948
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
Keywords: Decision making
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anecdotal Evidence (Active Comparator): Scenario describes a medication's (biologic's) therapeutic effect results based on anecdotal evidence.
  Interventions: Behavioral: Anecdotal Evidence
- Research Study Evidence (Active Comparator): Scenario describes a medication's (biologic's) therapeutic effect results based on research study evidence.
  Interventions: Behavioral: Research Study Evidence
- Anecdotal + Research Study Evidence (Active Comparator): Scenario describes a medication's (biologic's) therapeutic effect results based on research study evidence and anecdotal evidence.
  Interventions: Behavioral: Anecdotal + Research Study Evidence
- No Evidence (Placebo Comparator): Scenario describes a medication's (biologic's) therapeutic effect with no mention on anecdotal nor research study evidence.
  Interventions: Behavioral: No Evidence

INTERVENTIONS:
Behavioral: Anecdotal Evidence — Communicate basic information on the therapeutic effect of a drug using only anecdotal evidence.
  Arms: Anecdotal Evidence
Behavioral: Research Study Evidence — Communicate basic information on the therapeutic effect of a drug using only research study evidence.
  Arms: Research Study Evidence
Behavioral: Anecdotal + Research Study Evidence — Communicate basic information on the therapeutic effect of a drug using only anecdotal and research study evidence.
  Arms: Anecdotal + Research Study Evidence
Behavioral: No Evidence — Communicate basic information on the therapeutic effect of a drug using neither anecdotal evidence nor research study evidence.
  Arms: No Evidence

SUMMARY:
In dermatology, biologic medications are used to treat conditions such as moderate-to-severe psoriasis. These medications generally function to decrease inflammation or disrupt the inflammatory cycle. Examples of biologic medications commonly used in dermatology include tumor necrosis factor-alpha (TNF-alpha), blockers/inhibitors (etanercept, infliximab, certolizumab pegol, golimumab), interleukin 12/23 blockers (ustekinumab) and interleukin 17A blockers (secukinumab, ixekizumab).

Due to biologic medication's efficacy and safety profiles, they have revolutionized dermatology and the general medical field. However, patients may be apprehensive about choosing a biologic medication for a variety of reasons. These include hearing negative information about the drug from friends or family, being nervous about injection, or seeing the drug or its side effects negatively portrayed in the media. Many patients are not aware that clinical trial evidence for biologics exist, and instead may rely on anecdotal evidence in choosing to take these medications.

Because fear of the drug is inherently subjective, it can be modified with appropriate reassurance and presentation of evidence. Physicians must be able to ascertain from where the fear originates and how it can be countered. By understanding what kind of information will allow patients to be confident in their decision to take a biologic, dermatologists can improve outcomes and initiate use of this drug. Furthermore, reducing fear of side effects or adverse events may improve adherence to treatment and may improve treatment outcomes. The investigators propose this study with the goal of learning whether patients are more confident in the potential success of biologic medications in treating their psoriasis after being presented with clinical trial evidence, anecdotal evidence, or both.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with psoriasis (ICD-9: 696.1)
* Age 18-80

Exclusion Criteria:

* Individuals younger than 18 (line of questioning necessary for the study may be beyond understanding in this age group)
* Currently or previously managed with a biologic medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Oral survey responses | 1 day
  Oral survey response from 1 (not willing) to 10 (completely willing) scale to take a treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steve R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03168347/ICF_000.pdf